CLINICAL TRIAL: NCT00790348
Title: Effect of Januvia on Ghrelin and Other Gut Hormones in Patients With Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Berhane Seyoum, Wayne State University
Other Study IDs: 0709005250
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum of patients will be kept for future studies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients who on Januvia
- 2: Patients on Janumet (Combination of Januvia and Metformin)
- 3: Patients on Metformin

SUMMARY:
The purpose of this study is to see the effect of Januvia on Ghrelin levels in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes

Exclusion Criteria:

* Renal failure
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes on oral agent that require Metformin or Januvia only
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States